CLINICAL TRIAL: NCT01547312
Title: A Randomized Clinical Trial Using Fine Needle Aspiration For Evaluation of Hepatic Pharmacokinetics of MK-5172 in Participants With Chronic Hepatitis C
Brief Title: Evaluation of Hepatic Pharmacokinetics for Grazoprevir (MK-5172) in Participants With Chronic Hepatitis C (MK-5172-022)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 5172-022; 2011-004978-29 (EudraCT Number)
Record Dates: First submitted 2012-02-02; First posted 2012-03-07 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2b; Blood Specimen Collection; Ribavirin; grazoprevir

ARMS (4):
- Main Pt. 2: 800 mg Grazoprevir + Peg-IFN/RBV (Experimental): 800 mg Grazoprevir combined with Peg-Interferon/Ribavirin treatment.
  Interventions: Drug: Peg-Interferon; Procedure: Liver Samples from FNA; Procedure: Liver Samples from CNB; Procedure: Blood Samples; Drug: Ribavirin; Drug: 800 mg Grazoprevir
- Main Pt. 2: 100 mg Grazoprevir + Peg-IFN/RBV (Experimental): 100 mg Grazoprevir combined with Peg-Interferon/Ribavirin treatment.
  Interventions: Drug: Peg-Interferon; Procedure: Liver Samples from FNA; Procedure: Liver Samples from CNB; Procedure: Blood Samples; Drug: Ribavirin; Drug: 100 mg Grazoprevir
- Main Pt.1: 800 mg Grazoprevir (Experimental): 800 mg Grazoprevir.
  Interventions: Procedure: Liver Samples from FNA; Procedure: Liver Samples from CNB; Procedure: Blood Samples; Drug: 800 mg Grazoprevir
- Procedural Pilot (Experimental): Optimization of FNA procedure.
  Interventions: Procedure: Liver samples from CNB and FNA

INTERVENTIONS:
Drug: Peg-Interferon — Polyethyleneglycolated Interferon alfa-2b at 1.5 ug/kg/week, administered subcutaneously, once a week, over the entire course of the study.
  Other Names: PegIntron
  Arms: Main Pt. 2: 100 mg Grazoprevir + Peg-IFN/RBV; Main Pt. 2: 800 mg Grazoprevir + Peg-IFN/RBV
Procedure: Liver Samples from FNA — Tissue samples are collected at 3 separate visits, with each collection consisting of 3-4 fine needle aspiration (FNA) passes through the liver, guided by ultrasound.
  Arms: Main Pt. 2: 100 mg Grazoprevir + Peg-IFN/RBV; Main Pt. 2: 800 mg Grazoprevir + Peg-IFN/RBV; Main Pt.1: 800 mg Grazoprevir
Procedure: Liver Samples from CNB — Tissue samples are collected at 1 of six possible visits by core needle biopsy (CNB) of the liver.
  Arms: Main Pt. 2: 100 mg Grazoprevir + Peg-IFN/RBV; Main Pt. 2: 800 mg Grazoprevir + Peg-IFN/RBV; Main Pt.1: 800 mg Grazoprevir
Procedure: Blood Samples — Blood is collected from multiple blood draws, with the total volume for each participant not expected to exceed 500 ml.
  Arms: Main Pt. 2: 100 mg Grazoprevir + Peg-IFN/RBV; Main Pt. 2: 800 mg Grazoprevir + Peg-IFN/RBV; Main Pt.1: 800 mg Grazoprevir
Drug: Ribavirin — Ribavirin, 600-1400 mg administered orally, twice daily, over the entire course of the study.
  Other Names: Rebetol
  Arms: Main Pt. 2: 100 mg Grazoprevir + Peg-IFN/RBV; Main Pt. 2: 800 mg Grazoprevir + Peg-IFN/RBV
Drug: 800 mg Grazoprevir — 800 mg Grazoprevir administered orally, once per day, for 7 consecutive days.
  Arms: Main Pt. 2: 800 mg Grazoprevir + Peg-IFN/RBV; Main Pt.1: 800 mg Grazoprevir
Drug: 100 mg Grazoprevir — 100 mg Grazoprevir administered orally, once per day, for 7 consecutive days.
  Arms: Main Pt. 2: 100 mg Grazoprevir + Peg-IFN/RBV
Procedure: Liver samples from CNB and FNA — Tissue samples from the liver are collected by CNB as part of standard of care, and also by FNA during a single visit.
  Arms: Procedural Pilot

SUMMARY:
This study is divided into 2 segments, and proposes to qualify fine needle aspiration (FNA) as a platform to evaluate the hepatic pharmacokinetics of low and high oral doses of Grazoprevir (MK-5172) in non-cirrhotic participants chronically infected with hepatitis C virus (HCV). The first segment, is a procedural pilot conducted prior to the main study, that is aimed at ensuring optimal execution of the FNA procedure. During the procedural pilot, core needle biopsy (CNB) will be performed on participants as part of their standard of care, but no study drugs will be administered, nor will any procedures other than FNA be conducted. The second segment, the main study, is designed to evaluate the feasibility of measuring Grazoprevir by FNA. During the main study, drugs will be administered, and other additional procedures will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Has chronic compensated HCV infection.
* No contraindications to CNB or FNA procedures.
* Pilot study only: All comers with chronic HCV already scheduled to undergo CNB for fibrosis staging.
* Pilot study only: Requires a diagnostic liver biopsy to monitor progression of liver disease.
* Pilot study only: Does not have cirrhosis.
* Main study only: Males or non-pregnant and postmenopausal females willing to use medically acceptable contraception during, and for 6 months or longer after study.
* Main study only: Body mass index of 18.5 - 32.0 kg/m^2.
* Main study only: Can avoid aspirin, anticoagulants, and non steroidal inflammatory agents.
* Main study only: Has undergone prior treatment or is treatment naive for chronic HCV infection.

Exclusion Criteria for Main study only:

* History of any of the following: stroke, chronic seizures, major neurological disorders, gastric bypass surgery or bowel resection.
* No viral response to prior interferon based therapy.
* Prior treatment for HCV with an NS3/4A protease inhibitor.
* History of either clinically significant, uncontrolled endocrine, gastrointestinal, cardiovascular, hematological, immunological, renal, respiratory, or genitourinary abnormalities/diseases.
* History of neoplastic or myeloproliferative disease.
* Has any of the following : cirrhosis, decompensated liver disease, or other advanced liver disease, hepatocellular carcinoma, infection with human immunodeficiency virus (HIV), or hepatitis B.
* Evidence of high grade bridging fibrosis from prior liver biopsy or chronic hepatitis not caused by HCV.
* History of illicit drug use or alcohol abuse.
* Had surgery, donated at least one unit of blood, or participated in any other investigational study within 4 weeks prior to screening visit.
* History of multiple and/or severe allergies.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-05; Primary Completion 2012-11 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants from whom detectable concentrations of hepatic Grazoprevir are obtained by FNA. | Days 7-12.